CLINICAL TRIAL: NCT04602169
Title: Added Value of Superior Vena Cava Isolation in Patients With Pulmonary Vein Reconnection Undergoing Repeat Ablation for Recurrent Paroxysmal Atrial Fibrillation
Brief Title: Added Value of SVC Isolation in Patients With Pulmonary Vein Reconnection Undergoing Repeat Ablation for Recurrent Paroxysmal AF
Acronym: RECONNECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Sebastien Knecht, Professor Doctor, AZ Sint-Jan AV
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2721
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PVI only group (Active Comparator): Patients allocated to this group will receive PV re-isolation alone
  Interventions: Procedure: PVI
- PVI + SVC group (Active Comparator): Patients allocated to this group will receive PV re-isolation with SVC isolation.
  Interventions: Procedure: PVI + SVC

INTERVENTIONS:
Procedure: PVI — PV re-isolation will be conducted according to the CLOSE-protocol. Point-by-point radiofrequency (RF) delivery will be performed aiming for a contiguous circle enclosing all PVs. RF will be delivered in a power-controlled mode (without ramping) using 35-40 Watt. The irrigation rate will be set at 30 ml/min. RF will be delivered until an ablation index (AI) of ≥400 is reached at the posterior wall and ≥550 at the anterior wall. In case of dislocation, a new RF application reaching the AI target will be applied. Maximal intertag distance between two neighboring lesions is 6 mm. In case of intra-esophageal temperature (T°) rise >38.5°C during posterior LA wall ablation, RF delivery will stopped at an AI of 300. In the absence of first pass isolation, touch-up ablation was applied until PVI. In case of reconnection during the waiting time or during the adenosine test, the site of reconnection will be located and treated with touch-up ablation until adenosine proof PVI is reached.
  Arms: PVI only group
Procedure: PVI + SVC — Patients in this group receive PVI according to the CLOSE protocol. In addition, they will receive an SVC isolation. The circular mapping catheter will be introduced in the superior vena cava to determine baseline electrical activity and to confirm definite entrance and exit block after ablation. Ablation will be performed proximally to the SVC/right atrial junction with the contact force-catheter using circular point-by-point radiofrequency delivery with a power setting of 35W, targeting an AI ≥400. High output (25 mA) pacing will be applied before each RF application to check for phrenic nerve stimulation. In areas of phrenic nerve capture ablation will be avoided even in case of incomplete isolation.
  Arms: PVI + SVC group

SUMMARY:
Redo procedures after CLOSE-guided pulmonary vein isolation (PVI) for atrial fibrillation (AF) occur in 10% of patients. In case of pulmonary vein (PV) reconnection, electrophysiologists may re-isolate the pulmonary veins with or without the ablation of other commonly known PV-triggers. The superior vena cava (SVC) is one of the most common non PV-triggers for atrial tachyarrhythmias. SVC electrical isolation can be reached by circular radiofrequency-ablation under close monitoring of the phrenic nerve. However, it's added value remains unclear.

With this prospective, randomized, controlled, unblinded, mono-center study, the investigators aim to evaluate the 1-year recurrence rate in paroxysmal AF patients with reconnected pulmonary veins during a redo ablation with PV re-isolation or PV re-isolation with SVC isolation.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients scheduled for a repeat ablation of PAF after a previous PVI
* PV reconnection (in ≥1 PV's) found during procedure at the time of randomization

Exclusion Criteria:

* Patients with persistent AF
* Patients with durable PVI (no PVR)
* Previous ablation with isolation of the SVC, roofline, mitral line or previous vein of Marshal ethanol infusion
* Left atrial thrombus. LAA thrombus can be determined by preprocedural imaging: CT, TEE or MRI.
* Left ventricular ejection fraction <35%.
* Cardiac surgery within the previous 90 days.
* Expecting cardiac transplantation or other cardiac surgery within 180 days.
* Coronary PTCA/stenting within the previous 90 days or myocardial infarction within the previous 60 days.
* Documented history of a thromboembolic event within the previous 90 days.
* Diagnosed atrial myxoma.
* Significant restrictive, constrictive, or chronic obstructive pulmonary disease with chronic symptoms.
* Significant congenital anomaly or medical problem that in the opinion of the investigator would preclude enrollment
* Women who are pregnant or who plan to become pregnant between signing the informed consent form and the index ablation.
* Acute illness or active infection at time of index procedure
* Advanced renal insufficiency
* Unstable angina.
* History of blood clotting or bleeding abnormalities.
* Contraindication to anticoagulation.
* Life expectancy less than 1 year.
* Presence of a condition that precludes vascular access.
* INR greater than 3.5 within 24 hours of procedure - for patients taking warfarin.
* Patient cannot be removed from antiarrhythmic drugs for reasons other than AF.
* Unwilling or unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2020-11-16 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Recurrence of atrial tachyarrhythmia 1 year after the index ablation | 1 year after ablation
  Measured on 72hr Holter monitoring
Safety measured by procedural complications | From time of ablation to 1 month post procedure
  Occurence of procedural complications post procedure

SECONDARY OUTCOMES:
Total procedure time | At time of ablation
  Difference in total procedure time between groups
Fluoroscopy time | At time of ablation
  Difference in fluoroscopy time between groups
RF ablation time | At time of ablation
  Difference in RF ablation time between groups
Atrial volume | At time of ablation
  Evaluation of the atrial volume (ml)
SVC width | At time of ablation
  Evaluation of the SVC width (mm)
phrenic nerve width | At time of ablation
  Evaluation of the phrenic nerve width (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Sébastien Knecht, MD, PhD, Principal Investigator — AZ Sint-Jan AV
Locations (1):
- AZ Sint-Jan Brugge-Oostende AV, Bruges, Please Select, Belgium